CLINICAL TRIAL: NCT01521949
Title: A Phase 2 Study Acai Juice Product in Asymptomatic or Minimally Symptomatic Prostate Cancer Patients With Rising Prostate Specific Antigen (PSA)
Brief Title: Study of Acai Juice in Asymptomatic or Minimally Symptomatic Prostate Cancer Patients With Rising PSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0655.cc
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Nutraceutical; Acai Juice
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acai Juice (Experimental): 2 ounces of Acai Juice Product by mouth twice daily.
  Interventions: Drug: Acai Juice Product

INTERVENTIONS:
Drug: Acai Juice Product — 2 ounces of Acai Juice Product twice daily.
  Other Names: Acai Juice

SUMMARY:
Men who have Prostate Specific Antigen (PSA) recurrence with low PSA levels and long doubling times do not require immediate treatment with androgen deprivation therapy and may be safely observed. In these situations where current treatment options may cause more unnecessary side effects than anticipated benefit, it is reasonable to use a low-risk natural product such as Acai Juice Product with antioxidant properties to evaluate whether there are any anti-cancer effects.

DETAILED DESCRIPTION:
In this study, patients who meet eligibility criteria will take Acai Juice 2 ounces by mouth twice daily on a continuous basis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma.
* Evidence of rising PSA, on 2 separate occasions, at least one week apart.
* Baseline PSA must be ≥ 0.2 ng/mL at the time of screening. Radiographic evidence of disease is not required.
* Patients must have sufficient PSA time points prior to enrollment (a minimum of 3 PSA levels within a six month period) to calculate a baseline PSA doubling time.
* Patients may not be on active Luteinizing Hormone Releasing Hormone (LHRH) agonist therapy and must have testosterone level > 50 ng/dL.
* Patients must not be on active anti-androgen therapy or 5-alpha reductase inhibitors. However, patients who have been on a stable dose of 5-alpha reductase inhibitor for benign prostatic hypertrophy for at least 6 months may continue taking this agent.
* Patients who are on active surveillance for localized disease may participate in this study.
* Patients who are candidates for local salvage therapy must have had this option pursued or discussed; and the patient must have either declined salvage therapy or was deemed not to be a candidate for salvage therapy.
* Patients who have PSA recurrence after local salvage therapy may participate in this study.
* Patients with hormone sensitive disease who received prior androgen deprivation therapy as part of primary/salvage local treatment or patients receiving intermittent androgen deprivation therapy will be allowed to participate.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate hematologic function (absolute neutrophil count (ANC) ≥ 1,500 cells/µL; hemoglobin ≥ 9 g/dL, platelets ≥ 75,000/µL).
* Adequate renal function (serum creatinine ≤ 2 X the ULN).
* Adequate hepatic function (total bilirubin ≤ 2 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 3 x ULN, aspartate aminotransferase (AST) ≤ 3 x ULN).
* Agree not to take any other forms of natural or herbal supplements during study duration.
* Chemotherapy for prostate cancer is allowed as long as it was not given for hormone-refractory disease.

Exclusion Criteria:

* Inability to swallow liquids, or any medical condition that interferes with normal gastrointestinal absorption.
* Major surgery, radiation, or treatment with any other investigational drug within 2 weeks of study treatment.
* Documented hypersensitivity reaction to acai or any product contained in Acai Juice (see complete list in Appendix 1).
* Uncontrolled intercurrent disease (e.g. diabetes, hypertension, thyroid disease, coronary artery disease).
* Known chronic infection with human immunodeficiency virus (HIV) or viral hepatitis.
* Symptomatic prostate cancer as determined by cancer-related pain requiring narcotic pain medication.
* History of another cancer is exclusionary unless it is believed to be likely cured or is unlikely to be fatal in the next 3 years (e.g. squamous cell carcinoma, superficial bladder cancer, chronic lymphocytic leukemia, etc).
* Very fast PSA doubling time of less than 4 weeks, if the absolute PSA is > 2 ng/mL.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2013-12-25 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Lam, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of CO Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acai Juice
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acai Juice
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 69 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Gleason Score [Count of Participants; unit: Participants] — Gleason score is a system of grading prostate cancer tissue. A pathologist examines each biopsy core and determines a Gleason sum (X+Y=Z), ranging from 6 to 10. Gleason 6 cancers appear similar to normal prostate tissue and indicate that the tumor is less likely to spread and that have a low risk of recurrence after initial treatment. Gleason 8, 9, 10 cancers are high risk cancers, indicating that the tumor is more likely to spread and there is a high risk of cancer recurrence after initial treatment. Gleason 7 cancers are considered intermediate risk.
  Participants
    Gleason 6 (3+3) | 3
    Gleason 7 (3+4 or 4+3) | 14
    Gleason 8, 9, 10 (4+4, 4+5, 5+4, 5+5) | 4
Baseline PSA [Median (Full Range); unit: ng/dL] | 2.74 [0.33 to 43.4]

OUTCOME MEASURES:

1. Primary Outcome: PSA Response, as Defined by ≥ 50% Decrease in PSA From Baseline
Description: PSA will be obtained at baseline, every 6 weeks for the first 6 months, then every 3 months thereafter.
Time Frame: Two years
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Acai Juice
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Number of Participants With Increase in PSA Doubling Time in Comparison to Baseline
Description: Doubling time of PSA is the time that it takes for PSA to increase by 100%. Doubling time was calculated prior to starting study treatment and after starting study treatment.
Time Frame: Two years
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Acai Juice
Number analyzed (Participants) | 21
Participants | 15

ADVERSE EVENTS:
Time Frame: From study start through study completion, an average of 1 year.
Arm/Group | Acai Juice
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No